CLINICAL TRIAL: NCT04961567
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Litifilimab (BIIB059) in Adult Participants With Active Systemic Lupus Erythematosus Receiving Background Nonbiologic Lupus Standard of Care
Brief Title: A Study to Learn About the Safety of Litifilimab (BIIB059) Injections and Whether They Can Improve Symptoms of Adult Participants Who Have Systemic Lupus Erythematosus
Acronym: TOPAZ-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 230LE304; 2023-505696-74 (Other: EU CTIS)
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus; SLE; CLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Litifilimab High Dose (Experimental): Participants who are receiving background nonbiologic lupus SOC therapy will receive high dose of litifilimab, subcutaneously (SC), every 4 weeks (Q4W), up to Week 48 with an additional dose at Week 2.
  Interventions: Drug: Litifilimab
- Litifilimab Low Dose (Experimental): Participants who are receiving background nonbiologic lupus SOC therapy will receive low dose of litifilimab, SC Q4W, up to Week 48 with an additional dose at Week 2.
  Interventions: Drug: Litifilimab
- Placebo (Placebo Comparator): Participants who are receiving background nonbiologic lupus SOC therapy will receive litifilimab-matching placebo, SC Q4W, up to Week 48 with an additional dose at Week 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Litifilimab — Administered as specified in the treatment arm.
  Other Names: BIIB059
  Arms: Litifilimab High Dose; Litifilimab Low Dose
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
In this study, researchers will learn more about a study drug called litifilimab (BIIB059) in participants with systemic lupus erythematosus (SLE). The study will focus on participants who have active disease and are already taking standard of care medications. These may include antimalarials, steroids, and immunosuppressants.

The main objective of the study is to learn about the effect litifilimab has on lowering the activity of the disease. The main question researchers want to answer is:

- How many participants have an improvement in their symptoms after 52 weeks of treatment? Researchers will answer this and other questions by measuring the symptoms of SLE over time using a variety of scoring tools. These include the SLE Responder Index (SRI), the Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K), the British Isles Lupus Activity Group-2004 index (BILAG-2004), and the BILAG-BASED Combined Lupus Assessment (BICLA), among others.

Researchers will also learn more about the safety of litifilimab. They will study how participants' immune systems respond to litifilimab. Additionally, they will measure the effect litifilimab and SLE have on the quality of life of participants using a group of questionnaires.

The study will be done as follows:

* After screening, participants will be randomized to receive either a high or low dose of litifilimab, or placebo. A placebo looks like the study drug but contains no real medicine.
* All participants will receive either litifilimab or placebo as injections under the skin once every 4 weeks. The treatment period will last 52 weeks. Participants will continue to take their standard of care medications.
* Neither the researchers nor the participants will know if the participants are receiving litifilimab or placebo.
* There will be a follow-up safety period that lasts up to 24 weeks.
* In total, participants will have up to 22 study visits. The total study duration for participants will be up to 80 weeks.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate efficacy of litifilimab compared with placebo in participants with active SLE, who are receiving background lupus standard of care (SOC) therapy in reducing disease activity.

The secondary objectives of this study are to demonstrate efficacy of litifilimab compared with placebo in participants with active SLE, who are receiving background lupus SOC therapy in reducing disease activity and occurrence of flare up to Week 52; to demonstrate organ-specific efficacy of litifilimab compared with placebo in participants with active SLE, who are receiving background lupus SOC therapy in reducing joint disease activity and skin disease activity; to demonstrate and evaluate effect of litifilimab compared with placebo in reducing oral corticosteroid(s) (OCS) use; to evaluate additional efficacy of litifilimab compared with placebo in reducing disease activity with additional disease activity measures; assess the difference between litifilimab and placebo on participant reported health-related quality of life (HRQoL), symptoms, and impacts of SLE; to evaluate the safety, tolerability and immunogeneicty of litifilimab in participants with active SLE.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must be diagnosed with SLE at least 24 weeks prior to screening and must meet the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE, at screening by a qualified physician.
* Participant has a modified Systemic Lupus Erythematosus Disease Activity Index-200 (SLEDAI-2K) score ≥6 (excluding alopecia, fever, lupus-related headache, and organic brain syndrome) at screening (adjudicated).
* Participant has a modified clinical SLEDAI-2K score ≥4 (excluding anti-dsDNA, low complement component 3 [C3] and/or complement component 4 [C4], alopecia, fever, lupus-related headache, and organic brain syndrome) at screening (adjudicated) and randomization.
* Participant has BILAG-2004 grade A in ≥1 organ system or BILAG-2004 grade B in ≥2 organ systems at screening (adjudicated) and randomization.
* Participants must be treated with one of the following background nonbiologic lupus SOC therapies, initiated ≥12 weeks prior to screening and at stable dose ≥4 weeks prior to randomization:

  1. Antimalarials as stand-alone treatment
  2. Antimalarial treatment in combination with OCS and/or a single immunosuppressant
  3. Treatment with OCS and/or a single immunosuppressant.

Key Exclusion Criteria:

* History of or positive test result for human immunodeficiency virus (HIV).
* Current hepatitis C infection (defined as positive hepatitis C virus [HCV] antibody and detectable HCV ribonucleic acid [RNA]).
* Current hepatitis B infection (defined as positive for antibody to hepatitis B surface antigen [HBsAg] and/or positive for total antibody to hepatitis B core antigen [anti-HBc] with positive reflex HBV DNA).
* History of severe herpes infection.
* Presence of uncontrolled or New York Heart Association class III or IV congestive heart failure.
* Active severe lupus nephritis where, in the opinion of the investigator, protocol-specified SOC is insufficient and use of a more aggressive therapeutic approach, such as adding intravenous (IV) cyclophosphamide and/or high-dose IV pulse corticosteroid therapy or other treatments not permitted in the protocol, is indicated; or urine protein-creatinine ratio >2.0 or severe chronic kidney disease (estimated glomerular filtration rate <30 milliliters per minute per 1.73 meter square [mL/min/1.73 m^2]) calculated using the abbreviated Modification of Diet in Renal Disease equation.
* Any active skin conditions other than cutaneous lupus erythematosus (CLE) that may interfere with the study assessment of CLE such as but not limited to psoriasis, dermatomyositis, systemic sclerosis, non-LE skin lupus manifestation or drug-induced lupus.
* History or current diagnosis of a clinically significant non-SLE-related vasculitis syndrome.
* Active neuropsychiatric SLE.
* Use of oral prednisone (or equivalent) above 20 mg/day.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved a Systemic Lupus Erythematosus Responder Index of 4 (SRI-4) Response at Week 52 | Week 52
  An SRI-4 response is a composite endpoint defined by the following criteria:
  * Reduction from baseline of ≥4 points in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K).
  * No new organ system affected as defined by no new organ system with British Isles Lupus Assessment Group-2004 (BILAG-2004) grade A and no more than 1 new organ system with BILAG-2004 grade B compared with baseline.
  * No worsening from baseline in lupus disease activity as defined by <0.3-point increase on 3-point Physician's Global Assessment (PGA) - Visual Analog Scale (VAS).
  * No violation to protocol-specified medication rules.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved a British Isles Lupus Activity Group (BILAG) - Based Combined Lupus Assessment (BICLA) Response at Week 52 | Week 52
  The BILAG disease activity index evaluates SLE activity in number of organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows, BILAG A: severe disease activity; BILAG B: moderate disease activity; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved. BICLA is a composite endpoint defined as BILAG-2004 improvement, defined as all BILAG-2004 grade A at Baseline improved to grade B, C, or D, and all BILAG-2004 grade B at baseline improved to grade C or D, no BILAG-2004 worsening in other BILAG-2004 organ systems such that there are no new BILAG-2004 grade A or greater than 1 new BILAG-2004 grade B, no worsening in the SLEDAI-2K total score compared with Baseline, no worsening from Baseline in lupus disease activity defined by < 0.3-point increase on 3-point PGA-VAS and no violation to protocol-specified medication rules.
Percentage of Participants With at Least 4 Joints (Both Swollen and Tender) at Baseline Who Achieved a Joint-50 Response at Week 52 | Week 52
  Joint-50 response is 50% reduction in total active joint count from baseline. An active joint is defined as a joint with pain and signs of inflammation (e.g., tenderness, swelling or effusion). A 28-joint assessment will be performed to determine the active joint count, which is defined as the sum of tender and swollen joint counts.
Percentage of Participants With Oral Corticosteroid(s) (OCS) ≥10 milligrams per day (mg/day) at Baseline With OCS Reduction to ≤7.5 mg/day at Week 40, Which Is Sustained Through Week 52 With No Disease Worsening from Week 40 to Week 52 | Week 40 up to Week 52
  No worsening of the disease is defined as no new BILAG-2004 grade A or less than 2 new BILAG-2004 grade B since the last visit during the Week 40 to Week 52.
Percentage of Participants With a CLASI-A Score ≥10 at Baseline Who Achieved a 50% Improvement from Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity Score (CLASI-50) Response at Week 24 | Week 24
  Cutaneous Lupus Erythematosus Disease Area and Severity Index - Activity (CLASI-A) score is used to evaluate lupus skin manifestations. CLASI-A scores of 0 to 9, 10 to 20, and 21 to 70 represent disease severity of mild, moderate, and severe, respectively. CLASI-50 is 50% of improvement form baseline in CLASI-A.
Annualized Flare Rate Through Week 52 | Up to Week 52
  Annualized flare rate will be calculated as the total number of flares divided by the flare exposure time in days, and the ratio multiplied by 365.25.
Change from Baseline in Physician's Global Assessment (PGA) - Visual Analog Scale (VAS) Score by Visit | Up to Week 52
  The PGA is an investigator-administered assessment used to quantify disease activity and is measured using an anchored VAS. PGA asks the investigator to assess the participant's current disease activity from a score of 0 (none) to 3 (severe), with the assessment made relative to the most severe state of SLE.
Percentage of Participants Who Achieved a BICLA Response by Visit | Up to Week 52
  The BILAG disease activity index evaluates SLE activity in number of organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows, BILAG A: severe disease activity; BILAG B: moderate disease activity; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved. BICLA is a composite endpoint defined as BILAG-2004 improvement, defined as all BILAG-2004 grade A at Baseline improved to grade B, C, or D, and all BILAG-2004 grade B at baseline improved to grade C or D, no BILAG-2004 worsening in other BILAG-2004 organ systems such that there are no new BILAG-2004 grade A or greater than 1 new BILAG-2004 grade B, no worsening in the SLEDAI-2K total score compared with Baseline, no worsening from Baseline in lupus disease activity defined by < 0.3-point increase on 3-point PGA-VAS and no violation to protocol-specified medication rules.
Time to Onset of SRI-4 Response Sustained Through Week 52 | Up to Week 52
  An SRI-4 response is a composite endpoint defined by the following criteria:
  * Reduction from baseline of ≥4 points in SLEDAI-2K.
  * No new organ system affected as defined by no new organ system with BILAG-2004 grade A and no more than 1 new organ system with BILAG-2004 grade B compared with baseline.
  * No worsening from baseline in lupus disease activity as defined by <0.3-point increase on 3-point PGA-VAS.
  * No violation to protocol-specified medication rules.
Percentage of Participants Who Achieved SRI-4, -5, or -6 Response by Visit | Up to Week 52
  An SRI-4 response is a composite endpoint defined by the following criteria:
  * Reduction from baseline of ≥4 points in SLEDAI-2K.
  * No new organ system affected as defined by no new organ system with BILAG-2004 grade A and no more than 1 new organ system with BILAG-2004 grade B compared with baseline.
  * No worsening from baseline in lupus disease activity as defined by <0.3-point increase on 3-point PGA-VAS.
  * No violation to protocol-specified medication rules. SRI-5 and SRI-6 are computed with a minimal five-point or six-point improvement in SLEDAI-2K being required, respectively.
Percentage of Participants With Joint-50 Response by Visit | Up to Week 52
  Joint-50 response is 50% reduction in total active joint count from baseline. An active joint is defined as a joint with pain and signs of inflammation (e.g., tenderness, swelling or effusion). A 28-joint assessment will be performed to determine the active joint count, which is defined as the sum of tender and swollen joint counts.
Percentage of Participants With Baseline CLASI-A Score ≥10 Who Achieved a CLASI-20, -50, -70, or -90 Response by Visit | Up to Week 52
  Cutaneous Lupus Erythematosus Disease Area and Severity Index - Activity (CLASI-A) score is used to evaluate lupus skin manifestations. CLASI-A scores of 0 to 9, 10 to 20, and 21 to 70 represent disease severity of mild, moderate, and severe, respectively. CLASI-20, -50, -70 and -90 represent 20%, 50%, 70% or 90% improvement from baseline in CLASI-A score, respectively.
Percentage of Participants With Baseline CLASI-A Score ≥10 Who Achieved a CLASI-A Score of ≤1 by Visit | Up to Week 52
  Cutaneous Lupus Erythematosus Disease Area and Severity Index - Activity (CLASI-A) score is used to evaluate lupus skin manifestations. CLASI-A scores of 0 to 9, 10 to 20, and 21 to 70 represent disease severity of mild, moderate, and severe, respectively. CLASI-A ≤1 represent the absolute score ≤1 in CLASI-A by visit.
Percentage of Participants With Severe Flares Through Week 52 | Up to Week 52
  A SFI severe flare is defined any of the following:
  * Change in SLEDAI instrument score to >12.
  * New or worse: central nervous system SLE; vasculitis; nephritis; myositis; platelets <60,000 per milliliter (/mL); or hemolytic anemia with hemoglobin <7 grams per deciliter (g/dL) or decrease in hemoglobin >3 g/dL and requiring: doubling prednisone dose; or increase to >0.5 milligrams per kilogram per day (mg/kg/day) or hospitalization.
  * Increase in prednisone dose to >0.5 mg/kg/day.
  * New requirement for cyclophosphamide, azathioprine, methotrexate, or mycophenolate for SLE activity.
  * Hospitalization for SLE activity.
  * Increase in PGA score to >2.5
Time to First British Isles Lupus Activity Group-2004 (BILAG-2004) Severe Flare by Visit | Up to Week 52
  BILAG-2004 severe flare is defined as an A score for items recorded as worse or new. BILAG-2004 is evaluated by scoring each item of a list of signs and symptoms given as 4 = new; 3 = worse; 2 = same; 1 = improving; 0 = not present; and ND = not done.
Time to First Severe Flare as Defined by Safety of Estrogens in Systemic Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index Flare Index (SFI) | Up to Week 52
  SFI severe flare is defined any of the following: change in SLEDAI instrument score to >12; or new or worse: central nervous system SLE; vasculitis; nephritis; myositis; platelets <60,000 per milliliter (/mL); or hemolytic anemia with hemoglobin <7 grams per deciliter (g/dL) or decrease in hemoglobin >3 g/dL and requiring: doubling prednisone dose; or increase to >0.5 milligrams per kilogram per day (mg/kg/day) or hospitalization; or increase in prednisone dose to >0.5 mg/kg/day; or new requirement for cyclophosphamide, azathioprine, methotrexate, or mycophenolate for SLE activity; or hospitalization for SLE activity; or increase in PGA score to >2.5.
Percentage of Time Spent in Lupus Low Disease Activity State (LLDAS) | Up to Week 52
  LLDAS is a composite endpoint defined as:
  * SLEDAI-2K score ≤ 4, with no activity in a major organ system (renal, central nervous system, cardiopulmonary, vasculitis, fever); and
  * No new features of lupus disease activity compared with the previous assessment; and
  * Safety of Estrogens in Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) PGA ≤ 1; and
  * Current prednisone (or equivalent) dose ≤ 7.5 mg/day; and
  * Standard maintenance doses of immunosuppressive drugs and approved biological agents.
Percentage of Participants With Sustained LLDAS as Defined by the Number of Participants With ≥ 3, ≥ 5, and ≥ 7 Consecutive Visits in LLDAS up to and Including Week 52 | Up to Week 52
  LLDAS is a composite endpoint defined as:
  * SLEDAI-2K score ≤ 4, with no activity in a major organ system (renal, central nervous system, cardiopulmonary, vasculitis, fever); and
  * No new features of lupus disease activity compared with the previous assessment; and
  * SELENA-SLEDAI PGA ≤ 1; and
  * Current prednisone (or equivalent) dose ≤ 7.5 mg/day; and
  * Standard maintenance doses of immunosuppressive drugs and approved biological agents.
Percentage of Participants who Achieved LLDAS at Week 52 | Week 52
  LLDAS is a composite endpoint defined as:
  * SLEDAI-2K score ≤ 4, with no activity in a major organ system (renal, central nervous system, cardiopulmonary, vasculitis, fever); and
  * No new features of lupus disease activity compared with the previous assessment; and
  * SELENA-SLEDAI PGA ≤ 1; and
  * Current prednisone (or equivalent) dose ≤ 7.5 mg/day; and
  * Standard maintenance doses of immunosuppressive drugs and approved biological agents.
Percentage of Participants who Achieved SLEDAI-2K Improvement at Week 52 | Week 52
  The SLEDAI-2K is a reliable, valid, simple, 1-page activity index that measures disease activity and records features of active lupus as present or not. It uses a weighted checklist to assign a numeric score based on the presence or absence of 24 symptoms at the time of assessment or during the previous 28 days. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms), where higher scores represent increased disease activity. SLEDAI-2K improvement is defined as a reduction from Baseline of ≥ 4 points in SLEDAI-2K score.
Percentage of Participants who Achieved no Worsening of BILAG at Week 52 | Week 52
  The BILAG disease activity index evaluates SLE activity in number of organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows, BILAG A: severe disease activity; BILAG B: moderate disease activity; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved. No worsening of BILAG is defined as no new organ system affected, as defined by no new organ system with BILAG-2004 grade A and no more than 1 new organ system with BILAG-2004 grade B compared with Baseline.
Percentage of Participants who Achieved no Worsening of PGA-VAS at Week 52 | Week 52
  The PGA is an investigator-administered assessment used to quantify disease activity and is measured using an anchored VAS. PGA asks the investigator to assess the participant's current disease activity from a score of 0 (none) to 3 (severe), with the assessment made relative to the most severe state of SLE. No worsening from Baseline in lupus disease activity is defined by < 0.3-point increase on 3-point PGA-VAS.
Percentage of Participants who Achieved no Worsening of SLEDAI-2K at Week 52 | Week 52
  The SLEDAI-2K is a reliable, valid, simple, 1-page activity index that measures disease activity and records features of active lupus as present or not. It uses a weighted checklist to assign a numeric score based on the presence or absence of 24 symptoms at the time of assessment or during the previous 28 days. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms), where higher scores represent increased disease activity. No worsening of SLEDAI-2K is defined as no increase in the SLEDAI-2K total score from baseline.
Percentage of Participants who Achieved BILAG Improvement at Week 52 | Week 52
  The BILAG disease activity index evaluates SLE activity in number of organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows, BILAG A: severe disease activity; BILAG B: moderate disease activity; BILAG C: Stable mild disease; BILAG D: System previously affected but now inactive; BILAG E: System never involved. BILAG-2004 improvement, defined as all BILAG-2004 grade A at Baseline improved to grade B, C, or D, and all BILAG-2004 grade B at Baseline improved to grade C or D. BILAG-2004 improvement, defined as all BILAG-2004 grade A at Baseline improved to grade B, C, or D, and all BILAG-2004 grade B at Baseline improved to grade C or D. BILAG-2004 improvement, defined as all BILAG-2004 grade A at Baseline improved to grade B, C, or D, and all BILAG-2004 grade B at Baseline improved to grade C or D.
Percentage of Participants With OCS ≥ 10 mg/day at Baseline With OCS Reduction to ≤ 5 mg/day at Week 40, Which is Sustained Through Week 52 With no Disease Worsening From Week 40 to Week 52 | Week 40 up to Week 52
  No worsening of the disease is defined as no new BILAG-2004 grade A or less than 2 new BILAG-2004 grade B since the last visit between Week 40 and Week 52
Percentage of Participants With Baseline OCS ≥10 mg/day Who Achieved ≤7.5 mg/day at Week 52 | Week 52
Percentage of Participants With OCS ≥ 7.5 mg/day at Baseline With OCS Reduction to ≤ 7.5 mg/day at Week 52 | Week 52
Change from Baseline in Lupus-Specific Health-Related Quality-of-Life Questionnaire (LupusQoL) Score | Up to Week 52
  The LupusQoL is a participant-reported, lupus-specific, health-related quality-of-life questionnaire (HRQoL) consisting of 34 items grouped in 8 domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image and fatigue. Participants indicate their responses on a 5-point Likert response format, where 4 = never, 3 = occasionally, 2 = a good bit of the time, 1 = most of the time, and 0 = all the time. A LupusQoL score for each domain will be reported on a 0 to 100 scale, with greater values indicating better HRQoL.
Change from Baseline in Short Form Health Survey-36 (SF-36) Score | Up to Week 52
  SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary (PCS) score of SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement.
Change from Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score | Up to Week 52
  FACIT-Fatigue is a participant-administered HRQoL questionnaire that evaluates participant's fatigue in the 5 broad categories: physical well-being, social/family well-being, emotional well-being, functional well-being and additional concerns. The level of fatigue is measured by questions assessed on a 5-point scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The responses for each item are added to obtain a total score which ranges from 0 to 52, with a higher score indicating less fatigue.
Change from Baseline in Patient Health Questionnaire-9 (PHQ-9) Score | Up to Week 52
  PHQ-9 is a participant-administered HRQoL questionnaire to screen for the presence and severity of depression. The PHQ-9 is a participant-reported outcome (PRO) that is used to measure depression in adults. It contains 9 questions. The PHQ-9 yields an overall severity score that can range from 0 to 27 with the following severity scores: 0- 4 = none; 5-9 = mild; 10-14 = moderate; 15-19 = moderate-to-severe; and 20-27 = severe.
Change from Baseline in Work Productivity and Activity Impairment (WPAI): Lupus Score | Up to Week 52
  WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteeism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. Each score ranges from 0 to 100, with higher scores indicating greater impairment and less productivity.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to Week 52
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE is an AE that started or worsened in severity after the first dose of study treatment through 28 days after the last dose of study treatment or end of study (EOS) date, whichever comes earlier. An SAE is any untoward medical occurrence that at any dose results in death (a life-threatening event), in the view of the investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect, or is a medically important event.
Number of Participants With Antibodies to Litifilimab | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (177):
- United States (44):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Care Access Research - Huntington BeachCare Access Research - Huntington Beach, Huntington Beach, California
  - Valerius Medical Group, Los Alamitos, California
  - The Practice of Medicine, Los Angeles, California
  - R. Srinivasan, M.D., Inc. dba Monterey Park Medical Center, Monterey Park, California
  - Neurovations, Napa, California
  - Joo-Hyung Lee MD, Orange, California
  - Medvin Clinical Research, Whittier, California
  - RASF - Clinical Research Center, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Vida Clinical Research, Kissimmee, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - HMD Research, LLC, Orlando, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - The Emory Clinic Emory University, Atlanta, Georgia
  - Jefrey Lieberman, M.D., P.C., Decatur, Georgia
  - Southeastern Rheumatology Alliance dba Arthritis Center of North Georgia, Gainesville, Georgia
  - RNA America Health Sciences, Gainesville, Georgia
  - EBGS Clinical Trials, Snellville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Boston University School of Medicine, Boston, Massachusetts
  - DM Clinical Research - Boston, Brookline, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Saint Louis Rheumatology, St Louis, Missouri
  - Arthritis & Osteoporosis Associates, PA, Freehold, New Jersey
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - STAT Research, Dayton, Ohio
  - Piedmont Arthritis Clinic, P.A., Greenville, South Carolina
  - Low Country Rheumatology, PA, Summerville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Arthritis & Rheumatology Institute, Allen, Texas
  - Office of John P. Lavery M.D., PA, Allen, Texas
  - Tekton Research, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - R and H Clinical Research, Katy, Texas
  - Prime Clinical Research, Mansfield, Texas
  - SouthWest Rheumatology Research, LLC, Mesquite, Texas
  - Sun Research Institute, LLC, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
- Argentina (20):
  - Instituto de Investigaciones Clinicas Quilmes, Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, Buenos Aires, Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Policlìnica Red Omip S.A - Ensayos Clinicos GC, Mar del Plata, Buenos Aires
  - Centro Dermatologico Schejtman, San Miguel, Buenos Aires
  - APRILLUS Asistencia e Investigacion, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Instituto CAICI, Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Barrio Parque, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma Buenos Aires
  - STAT Research S.A., Ciudad Autonoma Buenos Aires
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro Privado de Medicina Familiar - Mind Out Research, Ciudad Autonoma Buenos Aires
  - Sanatorio Allende, Córdoba
  - Instituto de Reumatologia, Mendoza
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
- Belgium (2):
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
- Canada (3):
  - The Waterside Clinic, Barrie, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
- China (25):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The second Xiangya Hospital of Central South University, Changsha, Hu'nan
  - ZhuZhou Central Hospital, Zhuzhou, Hu'nan
  - EC of Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - Yanbian University Hospital (Yanbian Hospital), Yanji, Jilin
  - Jiujiang No.1 People's Hospital, Jiujiang, Jiujiang
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai, Shanghai Municipality
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
- Colombia (7):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Clínica de la Costa Ltda., Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas CIREEM S.A.S., Bogotá
  - Servimed S.A.S., Bucaramanga
  - IPS Centro Medico Julián Coronel S.A., Cali
  - Preventive Care Ltda, Chía
  - Healthy Medical Center, Zipaquirá
- Czechia (2):
  - Revmatologie s.r.o., Brno
  - Fakultni nemocnice Olomouc, Olomouc
- Germany (5):
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
- Hungary (5):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Bekes Varmegyei Kozponti Korhaz, Gyula
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt., Székesfehérvár
  - Vital Medical Center, Veszprém
- Israel (5):
  - Rambam Health Care Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale M. Scarlato, Scafati, Salerno
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedale-Università di Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Università Campus Bio-Medico di Roma, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
- Japan (33):
  - JCHO Chukyo Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - NHO Chibahigashi National Hospital, Chiba, Chiba
  - Chibaken Saiseikai Narashino Hospital, Narashino-shi, Chiba
  - KKR Hamanomachi Hospital, Fukuoka, Fukuoka
  - NHO Kyushu Medical Center, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Tonan Hospital, Sapporo, Hokkaido
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - NHO Osaka Minami Medical Center, Kawachinagano-shi, Osaka
  - Tazuke-kofukai Medical Research Institute Kitano Hospital, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Tokyo Medical and Dental University Hospital, Bunkyō City, Tokyo-To
  - St. Luke's International Hospital, Chūōku, Tokyo-To
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo-To
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo-To
  - Toho University Omori Medical Center, Ōta-ku, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo-To
- Netherlands (3):
  - Amsterdam UMC, Locatie VUMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - UMC Utrecht, Utrecht
- Centro Reumatologico, Caguas, Puerto Rico
- Romania (6):
  - S.C Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - S C Delta Health Care SRL, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - S.C.Centrul Medical Unirea SRL, Iași
  - Spitalul Judetean de Urgenta 'Sf. Ioan cel Nou' Suceava, Suceava
  - S.C Centrul Medical Unirea SRL, Târgu Mureş
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Bezanijska kosa, Belgrade
  - Institute of Treatment and Rehabilitation 'Niska Banja', Niška Banja
- United Kingdom (4):
  - Whipps Cross University Hospital, London, Greater London
  - Guy's Hospital, London, Greater London
  - Doncaster Royal Infirmary, Doncaster, South Yorkshire
  - Cannock Chase Hospital, Cannock, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- See also: Click here to learn more about this trial, visit our study website. — https://www.topazlupusstudy.com/